CLINICAL TRIAL: NCT01151592
Title: Assessment of Safety of Iron Sucrose (Venofer) in Patients With Chronic Kidney Disease Who Cannot Tolerate Ferumoxytol (Feraheme) or Iron Dextran (INFed or Dexferrum)
Brief Title: Safety Assessment of Iron Sucrose (Venofer) in Patients With Chronic Kidney Disease Who Cannot Tolerate Ferumoxytol (Feraheme) or Iron Dextran (INFed or Dexferrum)
Acronym: ASSURED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN10034
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia in Chronic Kidney Disease Patients
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iron Sucrose — Iron Sucrose, 1000 mg cumulative dose to be administered per the US package insert.
  Other Names: Venofer

SUMMARY:
The objective of this study is to assess the safety and tolerability of Venofer in patients with chronic kidney disease who cannot tolerate Ferumoxytol (Feraheme) or intravenous iron containing a dextran (INFed or Dexferrum).

DETAILED DESCRIPTION:
This is a Phase IV, multi-center, open label study that assesses the safety and tolerability of Iron Sucrose (Venofer) in subjects with CKD who require intravenous iron for the treatment of iron deficiency anemia (IDA) but cannot tolerate Ferumoxytol or Iron Dextran.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > or = to 18 years of age
* Determined by treating physician to have chronic kidney disease and require a course of intravenous iron
* Subject did not tolerate an intravenous iron containing a dextran or Ferumoxytol within the last year
* Subjects with hemodialysis-dependent or peritoneal dialysis chronic kidney disease should be receiving an erythropoiesis stimulating agent (ESA) as per the iron sucrose package insert

Exclusion Criteria:

* Known history of hypersensitivity or significant intolerance to iron sucrose
* Evidence of iron overload
* Hemochromatosis or other iron storage disorders
* Received an investigational drug within 30 days of screening
* Any other laboratory abnormality, medical condition or psychiatric disorder which would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements
* Pregnant or sexually-active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events, overall and related from Day of first iron sucrose administration through the end of the study. | Day 0 through 30 days after the final administration of iron sucrose

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States